CLINICAL TRIAL: NCT00329602
Title: A Parallel Group Study to Evaluate the Efficacy and Safety of Ropinirole for 26 Weeks and to Further Evaluate the Incidence of Augmentation and Rebound for a Further 40 Weeks Open-label Extension Treatment Period in Subjects Suffering From Moderate to Severe Restless Legs Syndrome.
Brief Title: Long-term Study Of Ropinirole In Restless Legs Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ROR104836
Record Dates: First submitted 2006-05-23; First posted 2006-05-25 (Estimated); Results first posted 2010-05-27 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Restless Legs Syndrome
Keywords: Moderate; Restless Legs Syndrome; Severe; ropinirole
MeSH Terms: conditions — Restless Legs Syndrome; Lymphoma, Follicular | interventions — ropinirole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Double-blind for 12 to 26 Weeks (Placebo Comparator): Double-blind (Ropinirole:Placebo) for 12 to 26 weeks
  Interventions: Drug: Placebo; Drug: Ropinirole
- Open-label ropinirole for 40-Weeks (Other): Open label ropinirole for 40 weeks
  Interventions: Drug: Ropinirole

INTERVENTIONS:
Drug: Placebo — Matching Placebo
  Arms: Double-blind for 12 to 26 Weeks
Drug: Ropinirole — Ropinirole IR 0.25mg/day to 4mg/day for RLS

SUMMARY:
This is an initial placebo-controlled study followed by open treatment evaluating the effectiveness and tolerability of ropinirole long-term in patients with moderate to severe Restless Legs Syndrome.

DETAILED DESCRIPTION:
A randomised, double-blind, placebo-controlled, parallel group study to evaluate the efficacy and safety of ropinirole for 26 weeks and to further evaluate the incidence of augmentation and rebound for a further 40 weeks open-label extension treatment period in subjects suffering from moderate to severe Restless Legs Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, between the ages of 18 and 79, inclusive

A female is eligible to enter and participate in the study if she is of:

1. Non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal); or,
2. Childbearing potential, has a negative result on all required pregnancy tests prior to randomisation, and agrees to an acceptable contraceptive method.

   * Subjects with a diagnosis of idiopathic RLS using the RLS Diagnostic Clinical Interview and the International RLS Study Group (IRLSSG) Diagnostic Criteria during the Screening Visit.
   * Subjects have had RLS symptoms with a history of a minimum of 15 RLS episodes during the previous month. If this is not possible due to the subject being on previous medication to treat RLS the investigator should ensure that the subject should have experienced 4-5 episodes of RLS symptoms during the last 7 days of the wash-out phase (see below). The subject must discontinue and wash-out any previous medication for the treatment of RLS or sleep prior to the Baseline Visit (Day 0). The minimum discontinuation period for wash-out is generally 5 half-lives of the medication or 7 consecutive evenings/nights medication-free prior to baseline, whichever is the longer period.
   * During the Wash-out and Screening Phase, RLS symptoms must be present for at least 4 of the last 7 nights immediately prior to the Baseline Visit (e.g., any combination of evenings and /or nights for = 4 days).
   * Subjects with a total score = 24 on the IRLS Rating Scale at baseline (Day 0).
   * Subjects with RLS symptoms that cause significant sleep impairment based on clinical judgment and guided by subject response to Question 4 of the IRLS Rating Scale (e.g., ordinarily this will include a response of (3) severe or (4) very severe sleep disturbance) at the Baseline Visit OR RLS symptoms that cause severe/very severe discomfort in the limbs based on clinical judgment and guided by subject response to Question 1 of the IRLS Rating Scale (e.g., this will include a response of (3) severe or (4) very severe discomfort in limbs) at the Baseline Visit (Day 0).
   * Subjects must be experiencing RLS symptoms requiring treatment at night-time.
   * Subjects must have given written informed consent prior to any specific study procedures.

Exclusion criteria:

* Subjects suffering from augmentation and/ or 'end of treatment' rebound RLS symptoms at baseline (Day 0). Augmentation is defined as RLS symptoms that occurred while on treatment and occur earlier in the afternoon/evening than they did before, symptoms which are more severe than when not treated, symptoms which start after less time at rest than they did before treatment, or symptoms which involve other parts of the body, such as the arms or trunk. 'End of treatment' rebound describes worsening of symptoms from baseline that occur after pharmacological treatment is stopped.
* Subjects with a previous history of augmentation.
* Subjects who have exhibited intolerance to ropinirole or any other dopamine agonist.
* Subjects requiring treatment of daytime RLS symptoms (daytime defined as 10:00 hours until 17:00 hours).
* Signs of secondary RLS (e.g., end stage renal disease, iron deficient anaemia or pregnancy at Baseline Visit).
* Subjects with a serum ferritin level of < 10 mcg/L (ng/mL) at Screening Visit.
* Subjects who suffer from a primary sleep disorder other than RLS that may significantly affect the symptoms of RLS (e.g. narcolepsy, sleep terror disorder, sleepwalking disorder, breathing related sleep disorder).
* Subjects diagnosed with movement disorders (e.g., Parkinson's Disease, dyskinesias, and dystonias).
* Subjects who have medical conditions which could affect efficacy assessments or clinically significant or unstable medical conditions that present a safety concern. These may include, but are not limited to, the following disorders: diabetes, peripheral neuropathy, rheumatoid arthritis, fibromyalgia syndrome, symptomatic orthostatic hypotension, severe cardiovascular disease, hepatic or renal failure, pleuro-pulmonary fibrosis, major psychotic illness.
* Subjects having a clinically significant abnormal laboratory value, ECG, or physical examination findings not resolved by the time of the baseline examinations (Day 0). Abnormal 12-lead ECG findings include, but are not limited to, the following: myocardial ischemia, clinically significant conduction abnormalities, or clinically significant arrhythmias.
* Subjects with a diastolic blood pressure = 110mmHg or = 50mmHg or systolic blood pressure = 180mmHg or = 90mmHg at the Screening or Baseline Visit.
* Subjects with a history of alcohol or substance abuse within the past year.
* Subjects taking any medication known to induce drowsiness, affect RLS or sleep and which have not been discontinued prior to the Baseline Visit. These medications include the following:

Atypical and typical antipsychotics, anticonvulsants, opioids (including propoxyphene and oxycodone), anxiolytics, all sedatives/hypnotics (including benzodiazepines), lithium, oral neuroleptics, stimulants (including methylphenidate), dopamine agonists (including ropinirole), dopamine antagonists (e.g., typical neuroleptics, metoclopramide), levodopa/carbidopa, clonidine, and sedating antihistamines (e.g., chlorpheniramine, diphenhydramine, hydroxyzine) or any preparations containing these antihistamines.

The minimum discontinuation period is generally 5 half lives or 7 consecutive evenings/nights medication free, prior to baseline, whichever is the longer period. Exceptions to this general rule are: fluoxetine, monoamine oxidase inhibitors: 4 weeks.

For subjects entering the 40-week, open-label treatment phase, the GSK Medical Monitor can be contacted to discuss individual cases where adherence to the above may not have occurred.

* Withdrawal, introduction, or change in dose of hormone replacement therapy (HRT) and/or any drug known to substantially inhibit CYP1A2 (e.g., ciprofloxacin, cimetidine, fluvoxamine, HRT) or induce CYP1A2 (e.g., tobacco, omeprazole) within 7 days prior to enrolment. Subjects already on these agents may be enrolled, but must remain on stable doses of the agents from 7 days prior to enrolment through to the follow-up visit at the end of the study.
* Night workers or any others whose sleeping habits are incompatible with the study design, or who would be required to make significant changes to their bedtime during the course of the study.
* Participation in any clinical drug or device trial in the one month prior to the Baseline Visit.
* Subjects who, in the opinion of the investigator, would be non-compliant with the visit schedules or other study procedures.
* Women who have a positive pregnancy test or who are lactating.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2006-03; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (37):
- Australia (5):
  - GSK Investigational Site, Camperdown, New South Wales
  - GSK Investigational Site, Kippa-Ring, Queensland
  - GSK Investigational Site, Woodville, South Australia
  - GSK Investigational Site, Clayton, Victoria
  - GSK Investigational Site, East Melbourne, Victoria
- Czechia (4):
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Ostrava
  - GSK Investigational Site, Pardubice
  - GSK Investigational Site, Prague
- Denmark (3):
  - GSK Investigational Site, Aalborg
  - GSK Investigational Site, Odense C
  - GSK Investigational Site, Vejle
- Germany (7):
  - GSK Investigational Site, Bamberg, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Regensburg, Bavaria
  - GSK Investigational Site, Marburg, Hesse
  - GSK Investigational Site, Westerstede, Lower Saxony
  - GSK Investigational Site, Schwerin, Mecklenburg-Vorpommern
  - GSK Investigational Site, Berlin, State of Berlin
- Italy (3):
  - GSK Investigational Site, Bologna, Emilia-Romagna
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Pavia, Lombardy
- GSK Investigational Site, Hamar, Norway
- Portugal (2):
  - GSK Investigational Site, Coimbra
  - GSK Investigational Site, Lisbon
- Slovakia (4):
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Dubnica nad Váhom
  - GSK Investigational Site, Levoča
  - GSK Investigational Site, Žilina
- Spain (3):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, San Sebastián
- Sweden (3):
  - GSK Investigational Site, Avesta
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Örebro
- Switzerland (2):
  - GSK Investigational Site, Bern
  - GSK Investigational Site, Zurich

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Garcia-Borreguero D, Hogl B, Ferini-Strambi L, Winkelman J, Hill-Zabala C, Asgharian A, Allen R. Systematic evaluation of augmentation during treatment with ropinirole in restless legs syndrome (Willis-Ekbom disease): results from a prospective, multicenter study over 66 weeks. Mov Disord. 2012 Feb;27(2):277-83. doi: 10.1002/mds.24889. Epub 2012 Jan 4. PMID 22328464
- [Derived] Giorgi L, Asgharian A, Hunter B. Ropinirole in patients with restless legs syndrome and baseline IRLS total scores >/= 24: efficacy and tolerability in a 26-week, double-blind, parallel-group, placebo-controlled study followed by a 40-week open-label extension. Clin Ther. 2013 Sep;35(9):1321-36. doi: 10.1016/j.clinthera.2013.06.016. Epub 2013 Aug 9. PMID 23938061
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: ROR104836 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: ROR104836 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: ROR104836 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: ROR104836 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: ROR104836 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: ROR104836 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: ROR104836 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (par.) could enter the Open-Label (OL) phase at the end of the Double-Blind (DB) phase. If a par. did not complete the DB phase due to lack of efficacy, he/she could also be considered for entry into the OL phase if the investigator considered it appropriate and the par. met the protocol-defined criteria in describing lack of efficacy.
Groups:
- Double-blind Placebo: Matching placebo tablets
- Double-blind Ropinirole IR: Ropinirole IR (immediate release) tablets containing ropinirole hydrochloride equivalent to 0.25 mg, 0.5 mg, 1.0 mg, or 2.0 mg of the active drug substance, taken once a day
- Open-label Ropinirole IR: Ropinirole IR (immediate release) tablets containing ropinirole hydrochloride equivalent to 0.5 mg, 1.0 mg, or 2.0 mg of the active drug substance, taken once a day
Period: 26-Week Double-Blind Treatment Phase
Arm/Group | Double-blind Placebo | Double-blind Ropinirole IR | Open-label Ropinirole IR
Started | 207 (Numbers of participants in the "Participant Flow" section are based on the Safety Population.) | 197 | 0
Completed | 88 | 98 | 0
Not Completed | 119 | 99 | 0
Not completed — Did not complete phase; reason unknown | 119 | 99 | 0
Period: 40-Week Open-Label Treatment Phase
Arm/Group | Double-blind Placebo | Double-blind Ropinirole IR | Open-label Ropinirole IR
Started | 0 | 0 | 269 (148 and 121 par. randomized to DB placebo and ropinirole IR, respectively, entered the OL phase.)
Completed | 0 | 0 | 233
Not Completed | 0 | 0 | 36
Not completed — Adverse Event | 0 | 0 | 20
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 2
Not completed — Lack of Efficacy | 0 | 0 | 9
Not completed — Captured as Other | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-Blind Placebo | Double-Blind Ropinirole IR | Total
Number analyzed (Participants) | 207 | 197 | 404
Age, Continuous [Mean (Standard Deviation); unit: years] — The Safety Population, comprised of all participants who received at least one dose of study medication, was used for all demographic characteristics.
  years | 55.9 (11.53) | 56.5 (11.97) | 56.2 (11.73)
Sex: Female, Male [Count of Participants; unit: Participants] — The Safety Population, comprised of all participants who received at least one dose of study medication, was used for all demographic characteristics.
  Participants
    Female | 132 | 124 | 256
    Male | 75 | 73 | 148
Race/Ethnicity, Customized [Number; unit: participants] — The Safety Population, comprised of all participants who received at least one dose of study medication, was used for all demographic characteristics.
  participants
    White | 204 | 197 | 401
    Asian | 2 | 0 | 2
    Hawaiian or other Pacific Islander | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in the International Restless Legs Syndrome (IRLS) Rating Scale Total Score at Week 12 and Week 26
Description: A 10-item, participant-reported scale covering different symptoms of the condition. Each item is scored from 0 to 4; 0 represents the absence of a problem and 4 reflects a very severe problem. The best and worst possible scores are 0 and 40, respectively; higher scores represent a greater severity of symptoms. A negative change from baseline indicates improvement, and a negative treatment difference indicates a benefit of Ropinirole IR over placebo. The primary assessment was made by calculating the difference in the average score obtained at Baseline with scores at Week 12 and then Week 26.
Time Frame: Baseline and Weeks 12 and 26
Population: Intention-to-Treat (ITT) Population: all randomised participants who received at least one dose of study medication, and for whom at least one valid post-baseline efficacy assessment was available. Analysis is based on the observed cases for each visit.
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Double-blind Placebo | Double-blind Ropinirole IR
Number analyzed (Participants) | 205 | 196
points on a scale
  Week 12, n=165, 164 | -12.1 (0.70) | -14.2 (0.71)
  Week 26, n=119, 123 | -13.4 (0.77) | -15.9 (0.76)
Statistical Analysis 1: Comparison: Double-blind Placebo vs Double-blind Ropinirole IR; Test type: Superiority or Other; p = 0.039, Repeated Measures Mixed Model — P-value is for Week 12; Adjusted for baseline IRLS Rating Scale total score, treatment group, visit, visit by treatment group interaction, and center group
Statistical Analysis 2: Comparison: Double-blind Placebo vs Double-blind Ropinirole IR; Test type: Superiority or Other; p = 0.023, Repeated Measures Mixed Model — P-value is for Week 26; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: Mean Change From Baseline in the International RLS (IRLS) Rating Scale Total Score at Weeks 1, 4, 8, 16, and 20
Description: A 10-item, participant-reported scale covering different RLS symptoms. Each item is scored from 0 to 4; 0 represents the absence of a problem and 4 reflects a very severe problem. The best and worst possible scores are 0 and 40, respectively; higher scores represent a greater severity of symptoms. The primary assessment from this study was made by calculating the difference in the average score obtained at Baseline with scores at Weeks 1, 4, 8, 16, and 20. Scores were adjusted for baseline IRLS total score, treatment group, visit, visit by treatment group interaction, and center group.
Time Frame: Baseline and Weeks 1, 4, 8, 16, and 20
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Double-blind Placebo | Double-blind Ropinirole IR
Number analyzed (Participants) | 205 | 196
points on a scale
  Week 1, n=198, 194 | -5.5 (0.52) | -7.8 (0.52)
  Week 4, n=183, 180 | -10.5 (0.60) | -13.6 (0.60)
  Week 8, n=168, 170 | -13.0 (0.66) | -15.3 (0.66)
  Week 16, n=137, 144 | -12.6 (0.75) | -15.0 (0.74)
  Week 20, n=125, 132 | -12.3 (0.78) | -15.7 (0.77)

3. Secondary Outcome: Change From Baseline in the Domains of the 12-item Medical Outcomes Study (MOS-12) Sleep Scale at Weeks 12 and 26
Description: The MOS-12 Sleep Scale is a comprehensive battery, which measures specific aspects of sleep in participants that may have varying co-morbidities, and, as a result, is appropriate for a medically diverse participant population. Domain values are presented on a 0-100 scale, where a higher score means a greater degree of the attribute implied by the scale name. Scores were adjusted for baseline MOS sleep scale domain value, treatment group, visit, visit by treatment interaction, and center group.
Time Frame: Baseline and Weeks 12 and 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Double-blind Placebo | Double-blind Ropinirole IR
Number analyzed (Participants) | 205 | 196
points on a scale
  Sleep disturbance, Week 12, n=153, 143 | -15.0 (1.62) | -24.0 (1.67)
  Sleep disturbance, Week 26, n=105, 97 | -16.4 (1.80) | -24.6 (1.87)
  Sleep adequacy, Week 12, n=153, 143 | 15.0 (1.91) | 22.8 (1.98)
  Sleep adequacy, Week 26, n=105, 97 | 14.9 (2.16) | 26.0 (2.25)
  Daytime somnolence, Week 12, n=153, 143 | -7.5 (1.28) | -11.4 (1.33)
  Daytime somnolence, Week 26, n=105, 97 | -9.1 (1.59) | -11.4 (1.65)

4. Secondary Outcome: Change From Baseline in Sleep Quantity, a Domain of the 12-item Medical Outcomes Study (MOS-12) Sleep Scale, at Weeks 12 and 26
Description: The MOS-12 Sleep Scale is a comprehensive battery, which measures specific aspects of sleep in participants that may have varying co-morbidities, and, as a result, is appropriate for a medically diverse participant population.Scores were adjusted for baseline MOS sleep scale domain value, treatment group, visit, visit by treatment interaction, and center group.
Time Frame: Baseline and Weeks 12 and 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Double-blind Placebo | Double-blind Ropinirole IR
Number analyzed (Participants) | 205 | 196
hours
  Week 12, n=153, 143 | 0.5 (0.10) | 0.7 (0.11)
  Week 26, n=105, 97 | 0.5 (0.11) | 0.7 (0.11)

5. Secondary Outcome: Change From Baseline in the Johns Hopkins RLS Quality of Life (RLS QoL) Questionnaire Overall Life Impact Score at Weeks 12 and 26
Description: The Johns Hopkins RLS QoL Questionnaire is a disease-specific instrument that assesses the impact of RLS on the daily life, emotional well-being, social life, and work life of participants. The overall life impact score for the John Hopkins RLS QoL scale ranges from a lowest possible score of 0 to a highest possible score of 100. Higher scores represent better quality of life. Scores were adjusted for baseline RLS Quality of Life score, treatment group, visit, visit by treatment interaction, and center group.
Time Frame: Baseline and Weeks 12 and 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Double-blind Placebo | Double-blind Ropinirole IR
Number analyzed (Participants) | 205 | 196
points on a scale
  Week 12, n=149, 141 | 14.0 (1.29) | 18.0 (1.33)
  Week 26, n=103, 94 | 16.5 (1.35) | 18.5 (1.41)

6. Secondary Outcome: Change From Baseline in the Domains of the MOS 36-item Short Form Health Survey (SF-36) at Weeks 12 and 26
Description: The MOS SF-36 is a generic QoL instrument measuring functional status and well-being. Positive change from baseline for all domains indicates improvement. For all MOS SF-36 domains, the minimum and maximum scores are 0 and 100, respectively, for the transformed scale. Scores were adjusted for baseline domain score, treatment group, visit, visit by treatment interaction, and center group.
Time Frame: Baseline and Weeks 12 and 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Double-blind Placebo | Double-blind Ropinirole IR
Number analyzed (Participants) | 205 | 196
points on a scale
  Bodily pain, Week 12, n=149, 142 | 12.3 (1.72) | 14.4 (1.76)
  Bodily pain, Week 26, n=104, 94 | 13.3 (2.01) | 14.0 (2.11)
  General health, Week 12, n=149, 142 | 3.0 (1.08) | 4.5 (1.11)
  General health, Week 26, n=104, 94 | 2.6 (1.31) | 4.1 (1.37)
  Mental health, Week 12, n=149, 142 | 5.0 (1.22) | 7.6 (1.26)
  Mental health, Week 26, n=104, 94 | 4.6 (1.25) | 6.2 (1.31)
  Physical functioning, Week 12, n=149, 142 | 2.4 (1.22) | 5.5 (1.25)
  Physical functioning, Week 26, n=104, 94 | 3.5 (1.48) | 2.6 (1.54)
  Role emotional, Week 12, n=149, 142 | 5.1 (1.62) | 7.0 (1.67)
  Role emotional, Week 26, n=104, 94 | 5.9 (1.66) | 6.6 (1.74)
  Role physical, Week 12, n=149, 142 | 5.2 (1.66) | 7.7 (1.71)
  Role physical, Week 26, n=104, 94 | 7.5 (1.85) | 6.7 (1.94)
  Social functioning, Week 12, n=149, 142 | 6.3 (1.58) | 9.8 (1.62)
  Social functioning, Week 26, n=104, 94 | 7.1 (1.56) | 8.8 (1.63)
  Vitality, Week 12, n=149, 142 | 8.0 (1.37) | 9.3 (1.41)
  Vitality, Week 26, n=104, 94 | 6.0 (1.54) | 9.2 (1.61)

7. Secondary Outcome: Percentage of Participants With a Score of Much/Very Much Improved on the Clinical Global Impression-Global Improvement (CGI-I) Scale at Weeks 1, 12 and 26
Description: The CGI-I is a psychometric instrument that is used to measure general clinical status in a variety of disease states. The CGI-I allows the investigator to rate the participant's global improvement or worsening compared with the condition at Baseline (Day 0). The scale is rated from 1-7 (1 = very much improved; 7 = very much worse). Typically, a participant with a score of 1 or 2 (much improved) is considered a responder.
Time Frame: Weeks 1, 12 and 26
Population: Intention-to-Treat (ITT) Population. Analysis is based on the observed cases for each visit.
Measure: Number; unit: percentage of participants
Arm/Group | Double-blind Placebo | Double-blind Ropinirole IR
Number analyzed (Participants) | 192 | 192
percentage of participants
  Week 1, n=192, 192 | 39 | 50
  Week 12, n=165, 160 | 86 | 109
  Week 26, n=112, 108 | 72 | 91

8. Secondary Outcome: Number of Participants Withdrawing Due to Lack of Efficacy During the First 26 Weeks of the Study
Description: Lack of efficacy is defined as up to a 10% improvement in the IRLS Rating Scale total score from the participant's Baseline value and at least 12 weeks of treatment during the double-blind phase.
Time Frame: Baseline to Week 26
Population: Intention-to-Treat (ITT) Population: all randomised participants who received at least one dose of study medication, and for whom at least one valid post-baseline efficacy assessment was available
Measure: Number; unit: participants
Arm/Group | Double-blind Placebo | Double-blind Ropinirole IR
Number analyzed (Participants) | 205 | 196
participants | 2 | 3

9. Secondary Outcome: Number of Participants Rated as Normal or Borderline Ill on the CGI Severity of Illness (CGI-S) Scale at Week 26
Description: The CGI-S scale is a psychometric instrument that is used to measure general clinical status in a variety of disease states. The CGI-S allows the investigator to rate the severity of the participant's illness considering their total clinical experience with the subject population being studied and on all information available at the time of rating. The scale is rated from 1-7 (1 = normal, not at all ill; 2 = borderline ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severly ill; 7 = among the most extremely ill participants).
Time Frame: Week 26
Population: Intention-to-Treat (ITT) Population: all randomised participants who received at least one dose of study medication, and for whom at least one valid post-baseline efficacy assessment was available. Data are presented for the participants still in the study and assessed at Week 26, which is less than those randomised at baseline.
Measure: Number; unit: participants
Arm/Group | Double-blind Placebo | Double-blind Ropinirole IR
Number analyzed (Participants) | 112 | 108
participants | 50 | 50

10. Secondary Outcome: Median Time to First CGI-I Response of Much/Very Much Improved During the Double-blind Phase
Description: The median time to first CGI-I response of much/very much improved was calculated. The CGI-I is a psychometric instrument that is used to measure general clinical status in a variety of disease states. The CGI-I allows the investigator to rate the participant's global improvement or worsening compared with the condition at Baseline (Day 0). The scale is rated from 1-7 (1 = very much improved; 7 = very much worse). Typically, a participant with a score of 1 or 2 (much improved) is considered a responder.
Time Frame: Baseline to Week 26
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Double-blind Placebo | Double-blind Ropinirole IR
Number analyzed (Participants) | 205 | 196
days | 28 [22 to 33] | 21 [14 to 21]

11. Secondary Outcome: Number of Participants With a Score of Much/Very Much Improved on the CGI-I Scale at Week 67
Description: as for outcome 7
Time Frame: Week 67
Population: Open-Label (OL) ITT Population: all participants who were enrolled into the OL Phase of the study, received at least one dose of OL study medication, and had a baseline IRLS total score and on-treatment IRLS assessment. Data are presented for participants still in the study and assessed at Week 26, which is less than those randomized at baseline.
Measure: Number; unit: participants
Arm/Group | Open-label Ropinirole IR
Number analyzed (Participants) | 200
participants | 184

12. Primary Outcome: Number of Participants With Clinically Meaningful Augmentation and Early Morning Rebound (EMR) Cases
Description: Clinically meaningful augmentation and early morning rebound (EMR) were assessed and confirmed by an independent Adjudication Board. EMR describes the development of RLS symptoms during the early morning, following therapeutic intervention. EMR is differentiated from augmentation, in which the earlier onset of symptoms occurs in the evening.
Time Frame: During 15-month study duration at scheduled (Weeks 16, 20, 26, or early withdrawal for DB phase; Weeks 39, 47, 55, 63, 67, or early withdrawal for the OL phase) and unscheduled (26-week DB phase and 40-week OL phase) visits
Population: Safety Population: all participants who received at least one dose of study medication
Measure: Number; unit: participants
Arm/Group | Overall Study | Double-blind Placebo | Double-blind Ropinirole IR | Open-label Ropinirole IR
Number analyzed (Participants) | 404 | 207 | 197 | 269
participants
  Confirmed augmentation | 15 | 1 | 7 | 8
  Clinically meaningful augmentation | 11 | 1 | 5 | 5
  Confirmed EMR | 7 | 1 | 4 | 2

13. Secondary Outcome: Mean Change From Baseline in the IRLS Rating Scale Total Score at Week 67
Description: A 10-item, participant-reported scale covering different symptoms of the condition. Each item is scored from 0 to 4, with 0 representing the absence of a problem and 4 reflecting a very severe problem. The best and worst possible scores are 0 and 40, respectively. The primary assessment was made by calculating the difference in the average score obtained at Baseline with score at Week 67.
Time Frame: Baseline and Week 67
Population: Open-Label ITT Population: all participants who were enrolled into the Open-Label Phase of the study, received at least one dose of Open-Label study medication, and had a baseline IRLS total score and on-treatment IRLS assessment. Analysis is based on the observed cases for each visit.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Open-label Ropinirole IR
Number analyzed (Participants) | 268
points on a scale | -20.4 (8.36)

14. Post Hoc Outcome: Post-hoc Analysis of Mean Change From Baseline in the International Restless Legs Syndrome (IRLS) Rating Scale Total Score at Week 12 and Week 26, Exploring the Impact of Center Group on Treatment Effect
Description: A post-hoc analysis of the primary outcome measure, exploring the variation in treatment effects across center groups by excluding those with the most extreme treatment effects, was conducted. Centers were grouped into five center groups.
Time Frame: Baseline and Weeks 12 and 26
Population: ITT Population excluding the two center groups with the most extreme treatment effects. Analysis is based on the observed cases for each visit.
Measure: Least Squares Mean (Standard Error); unit: Points on a scale
Groups:
- Double-blind Placebo: Double-Blind Placebo participants (receiving matching placebo tablets) who were not in the center groups with the highest or lowest treatment effects
- Double-blind Ropinirole IR: Double-Blind Ropinirole participants (receiving Ropinirole IR [immediate release] tablets containing ropinirole hydrochloride equivalent to 0.25 mg, 0.5 mg, 1.0 mg, or 2.0 mg of the active drug substance, taken once a day) who were not in the center groups with the highest or lowest treatment effects
Arm/Group | Double-blind Placebo | Double-blind Ropinirole IR
Number analyzed (Participants) | 136 | 134
Points on a scale
  Week 12, n=136, 134 | -12.2 (0.78) | -13.8 (0.79)
  Week 26, n=103, 105 | -14.0 (0.84) | -15.7 (0.83)

15. Post Hoc Outcome: Post-hoc Analysis of Percentage of Participants With a Score of Much/Very Much Improved on the Clinical Global Impression-Global Improvement (CGI-I) Scale at Weeks 12 and 26, Exploring the Impact of Center Group on Treatment Effect
Description: A post-hoc analysis of CGI-I, exploring the variation in treatment effects across center groups by excluding the same two center groups as in the IRLS post-hoc analysis, was conducted. Centers were grouped into five center groups.
Time Frame: Weeks 12 and 26
Population: ITT Population excluding the same two center groups as in the IRLS post-hoc analysis. Analysis is based on the observed cases for each visit.
Measure: Number; unit: Number of responders
Groups:
- Double-blind Placebo: Double-Blind Placebo participants (receiving matching placebo tablets) who were not excluded from the IRLS post-hoc analysis
- Double-blind Ropinirole IR: Double-Blind Ropinirole participants (receiving Ropinirole IR [immediate release] tablets containing ropinirole hydrochloride equivalent to 0.25 mg, 0.5 mg, 1.0 mg, or 2.0 mg of the active drug substance, taken once a day) who were not excluded from the IRLS post-hoc analysis
Arm/Group | Double-blind Placebo | Double-blind Ropinirole IR
Number analyzed (Participants) | 136 | 134
Number of responders
  Week 12, n=136, 134 | 75 | 93
  Week 26, n=99, 96 | 63 | 82

ADVERSE EVENTS:
Arm/Group | Double-blind Placebo | Double-blind Ropinirole IR | Open-Label Ropinirole IR
Serious Adverse Events (participants affected / at risk) | 6/207 | 6/197 | 11/269
Other Adverse Events (participants affected / at risk) | 71/207 | 123/197 | 122/269
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Placebo (N=207) | Double-blind Ropinirole IR (N=197) | Open-Label Ropinirole IR (N=269)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Fallopian tube cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Ovarian cyst torsion (Reproductive system and breast disorders) | 1 | 0 | 0
Gallbladder disorder (Hepatobiliary disorders) | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Bursa calcification (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Brain stem ischaemia (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Placebo (N=207) | Double-blind Ropinirole IR (N=197) | Open-Label Ropinirole IR (N=269)
Nausea (Gastrointestinal disorders) | 16 | 83 | 67
Headache (Nervous system disorders) | 23 | 29 | 20
Fatigue (General disorders) | 14 | 28 | 29
Nasopharyngitis (Infections and infestations) | 14 | 21 | 33
Dizziness (Nervous system disorders) | 6 | 20 | 16
Vomiting (Gastrointestinal disorders) | 0 | 22 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 7 | 9
Insomnia (Psychiatric disorders) | 5 | 12 | 1
Diarrhea (Gastrointestinal disorders) | 5 | 10 | 3
Somnolence (Nervous system disorders) | 4 | 9 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.